CLINICAL TRIAL: NCT00569153
Title: A Phase 1/2, Open-Label, Multiple-Dose Study of the Safety, Tolerability, and Pharmacokinetics of TAK-700 in Metastatic, Androgen-Independent Prostate Cancer Subjects
Brief Title: Safety Study of TAK-700 in Subjects With Prostate Cancer.
Acronym: TAK-700
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-700_201; TAK-700-201
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Prostatic Neoplasms
Keywords: Androgen-independent prostate cancer, metastatic
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — orteronel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (TAK-700) (Experimental)
  Interventions: Drug: TAK-700
- Arm 2 (TAK-700 at 400 mg & 5 mg prednisone) (Experimental)
  Interventions: Drug: TAK-700
- Arm 3 (TAK-700 at 600 mg & 5 mg prednisone) (Experimental)
  Interventions: Drug: TAK-700
- Arm 4 (TAK-700 at 600 mg) (Experimental)
  Interventions: Drug: TAK-700

INTERVENTIONS:
Drug: TAK-700 — Phase 1 portion of study:
  TAK-700 dose escalation. Tablets administered orally, twice daily until disease progression or occurrence of an unacceptable adverse event.
  Phase 2 portion of study:
  Patients will receive one of 4 treatments:
  * TAK-700 at 300 mg twice/day
  * TAK-700 at 400 mg and 5 mg prednisone twice/day
  * TAK-700 at 600 mg and 5 mg prednisone twice/day
  * TAK-700 at 600 mg once/day in the morning

SUMMARY:
The purpose of this study is to determine the safety and tolerability of TAK-700 in patients with asymptomatic metastatic, androgen independent prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male and at least 18 years of age.
* Subject has histologically- or cytologically-confirmed prostate adenocarcinoma with metastatic, progressive disease while on androgen deprivation therapy.
* Subject has radiograph-documented (computed tomography, magnetic resonance imaging or x-ray) metastatic disease.
* Subject has undergone orchiectomy or is expected to continue receiving luteinizing hormone-releasing hormone analogue therapy, and has a testosterone level of <50 ng/dL at screening.
* Subject has discontinued all antiandrogen therapy (within 30 days for flutamide and within 6 weeks for all others) prior to their first dose of study drug.
* Subject has a prostate-specific antigen level ≥5 ng/mL.
* Subject meets all screening laboratory values as specified in the protocol.
* Subject has a screening ejection fraction that is above the lower limit of the institutional normal range.
* Subject has ECOG performance status of 0 to 2.
* Subject has normal or, in the opinion of the investigator, clinically insignificant, physical examination findings, ECG and chest x-ray results.
* Subjects, even if surgically sterilized (ie, status postvasectomy), who: agree to practice effective barrier contraception during the entire study treatment period and for 4 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourse.

Exclusion Criteria:

* Subject has known hypersensitivity to TAK-700 or related compounds.
* Subject has received prior therapy with aminoglutethimide or ketoconazole within 30 days prior to the first dose of study drug.
* Subject has received prior chemotherapy for prostate cancer.
* Subject has received any investigational compound within 30 days prior to first dose of study drug.
* Subject has received prior herbal product known to decrease prostate-specific antigen levels (eg, Saw Palmetto, PC-SPES) within 30 days prior to the first dose of study drug.
* Subject has received radiation therapy for prostate cancer within 30 days prior to first dose of study drug.
* Chronic therapy with oral or other systemically administered corticosteroids, such as prednisone, within 30 days prior to Screening. Chronic therapy is defined as the use of corticosteroids for more than 7 days within a 30-day period.
* Subject has current spinal cord compression, current bilateral hydronephrosis, or current bladder neck outlet obstruction.
* Subject has a history of adrenal insufficiency.
* Subject has a history of myocardial infarction, ischaemic symptomatic heart disease, cardiac arrhythmias or thromboembolic events (eg, deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular events), or any other cardiac condition (e.g., pericardial effusion restrictive cardiomyopathy) within 12 months prior to first dose of study drug.
* Subject has any symptoms which the investigator deems related to prostate cancer, i.e., bone pain, pelvic pain.
* Subject has a history of congestive heart failure (New York Heart Association Class II or greater.
* Subject has history of another malignancy other than basal cell carcinoma or state 1 squamous cell carcinoma of the skin, within the last 5 years.
* Subject has uncontrolled hypertension.
* Subject is known to have HIV infection, chronic Hepatitis B or C or any other serious medical condition or psychiatric illness that might affect life expectancy or make it difficult to successfully manage and follow the subject according to protocol.
* Subject is unable to understand verbal or written English or any other language for which a certified translation of the institutional review board (IRB)-approved informed consent has been provided.
* Subject is unwilling or unable to comply with the protocol or cooperate fully with the investigator and site personnel.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2008-04; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of TAK-700 by evaluating adverse events, vital signs, physical examination findings, concomitant medications and laboratory tests. | Cycle 1: Weeks 1, 2, 3 and 4, then every 4 weeks thereafter.

SECONDARY OUTCOMES:
Efficacy and pharmacokinetics (PSA response and/or objective disease response) | Cycle 1: Weeks 1, 2, 3 and 4, then every 4 weeks thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (19):
- United States (19):
  - USC Westside Prostate Cancer Center, Beverly Hills, California
  - University of Southern California, Los Angeles, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - South Florida Medical Research, Aventura, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Northwestern University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Chicago Pharmacy, Chicago, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Kellogg Pharmacy - Evanston Hospital, Evanston, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Kellogg Cancer Care Center, Glenview, Illinois
  - Hematology/Oncology Associates of Central New York, East Syracuse, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Taussig Cancer Institute, Cleveland, Ohio
  - Tennessee Oncology, Nashville, Tennessee